CLINICAL TRIAL: NCT02497820
Title: A Randomised Double Blind Dose Non-inferiority Trial of a Daily Dose of 600mg Versus 300mg Versus 100mg of Enteric Coated Aspirin as a Cancer Preventive in Carriers of a Germline Pathological Mismatch Repair Gene Defect, Lynch Syndrome
Brief Title: Finding the Best Dose of Aspirin to Prevent Lynch Syndrome Cancers
Acronym: CaPP3 Israel
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Rambam Health Care Campus (Other); Rabin Medical Center (Other); Soroka University Medical Center (Other); Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0246-14-TLV
Record Dates: First submitted 2015-07-07; First posted 2015-07-15 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Lynch Syndrome I (Site-specific Colonic Cancer)
MeSH Terms: conditions — Lynch syndrome I (site-specific colonic cancer) | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 100 mg daily aspirin (Active Comparator): They will receive one small tablets each day for two years in a blinded fashion
  Interventions: Drug: Aspirin
- 300 mg daily aspirin (Active Comparator): They will receive two large enteric coated tablets each day for two years in a blinded fashion
  Interventions: Drug: Aspirin
- 600 mg daily aspirin (Active Comparator): They will receive two large enteric coated tablets each day for two years in a blinded fashion
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Aspirin (acetylsalicylic acid) has a marketing approval for use in the EU and is widely available as an over the counter medicine. However it is not being used within its licensed indication and the aspirin (at any dose in this study) will be treated as an investigational medicinal product (IMP).
  Tablets will be provided as enteric-coated 100mg or 300mg tablets for oral use. All patients will receive at least some dose of aspirin but blinding to the actual dose will be achieved by the use of 'dummy' tablets using the same excipients as in the active formulation of the aspirin minus the active ingredient.
  The aspirin and dummy tablets should be stored at room temperature below 25⁰C in a dry place.
  Other Names: acetylsalicylic acid

SUMMARY:
A randomised double blind dose non-inferiority trial of a daily dose of 600mg versus 300mg versus 100mg of enteric coated aspirin as a cancer preventive in carriers of a germline pathological mismatch repair gene defect, Lynch Syndrome. Project 3 in the Cancer Prevention Programme (CaPP3).

DETAILED DESCRIPTION:
Study design: A randomised, double-blind, dose non-inferiority study.

Study Intervention: Enteric-coated aspirin 100mg, 300mg or 600mg blinded dose daily followed by daily 100mg open label dose daily.

Primary objective: To determine whether the cancer preventive properties of enteric coated aspirin in Lynch syndrome are dose sensitive by comparing overall cumulative Lynch syndrome cancer incidence rates after 5 years in people who took 100mg, 300mg or 600mg enteric coated aspirin for at least 2 years.

Secondary objectives: Compare overall cumulative incidence of primary colorectal cancers using Poisson regression to allow for multiple primaries in individual patients in the three treatment groups.

Compare overall cumulative incidence of primary endometrial cancers using Poisson regression to allow for multiple primaries in individual patients in the three treatment groups.

Compare overall cumulative incidence of cancers of all types, using Poisson regression to allow for multiple primaries in individual patients in the three treatment groups.

The burden of adverse events associated with the different aspirin doses in this relatively young and healthy population will be documented.

Primary outcome: The number of new primary mismatch repair deficient cancers ("Lynch syndrome cancers") at 5 years and beyond which develop in participants who remain on prescribed treatment for a minimum of 2 years.

Number of study sites: 4 ISRAEL sites. 20 sites all over the world.

Study population/size: 300 patients in ISRAEL. UK 1000-1500 patients. Total with International 3,000 patients.

Study duration: 7 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years.
2. Confirmed germline pathological variant in one of the mismatch repair genes; MSH2, MLH1, PMS2 or MSH6 or a 3' EPCAM deletion associated with MSH2 silencing or be a carriers of a constitutional epimutation manifesting a classic Lynch syndrome phenotype.
3. Able to swallow tablets.
4. Provision of voluntary written informed consent.

Exclusion Criteria:

1. Regular use of a non-steroidal anti-inflammatory agent (except aspirin*) on a prescription and/or long-term basis. Regular is defined as > 3 doses per week.
2. Regular use of aspirin (> 3 doses per week or on a prescription basis) that cannot be replaced with any one of the randomised arms of the study followed by 100mg dose.
3. Current methotrexate use at a weekly dose of ≥ 15mg.
4. Known aspirin intolerance or hypersensitivity, including aspirin-sensitive asthma.
5. Existing clinically significant liver impairment.
6. Existing renal failure.
7. Confirmed active peptic ulcer disease within the previous three months.
8. Known bleeding diathesis or concomitant warfarin therapy.
9. Inability to comply with study procedures and agents.
10. Women reporting that they are pregnant or actively planning to achieve a pregnancy within the next two years.
11. Women who are breastfeeding.
12. Any significant medical illness that would interfere with study participation.

    * Previous use of aspirin for medicinal purposes does not exclude enrolment but duration and quantity need to be documented in detail

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2016-09; Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
cancer preventive properties of enteric coated aspirin in Lynch syndrome are dose sensitive by comparing overall cumulative Lynch syndrome cancer | 5 years
  The number of new primary mismatch repair deficient cancers ("Lynch syndrome cancers") at 5 years which develop in participants who remain on prescribed treatment for a minimum of 2 years.

SECONDARY OUTCOMES:
Overall cumulative of new colorectal cancers incidence rates after 5 years | 5 years
  The number of new colorectal cancers at 5 years which develop in participants who remain on prescribed treatment for a minimum of 2 years.
Overall cumulative of new endometrial cancers incidence rates after 5 years | 5 years
  The number of new endometrial cancers at 5 years which develop in participants who remain on prescribed treatment for a minimum of 2 years.
Overall cumulative of new new cancers of all types incidence rates after 5 years | 5 years
  • The number of new cancers of all types at 5 years which develop in participants who remain on prescribed treatment for a minimum of 2 years.
Overall cumulative of changes in the titre of frameshift peptide antibodies after 2 & 5 years | 5 years
  Changes at 2 & 5 years in the titre of frameshift peptide antibodies from commencement of the prescribed treatment.
Overall cumulative of of new adenomas at five years | 5 years
  The number of new adenomas at five years

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Arber, MD, MSc, MHA, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel